CLINICAL TRIAL: NCT02749084
Title: Multiple Donor Regulatory T Cell (Treg) Infusions (T Reg DLI) for Severe Refractory Chronic Graft Versus Host Disease (GVHD) After Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Multiple Donor Treg DLI for Severe Refractory Chronic GVHD
Acronym: TREG2015001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mario Arpinati (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor-Investigator, Mario Arpinati, Dr Mario Arpinati, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Organization: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160/2015/O/Sper
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Chronic Graft Versus Host Disease
Keywords: chronic graft versus host disease; T regulatory cell
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- T reg DLI (Experimental): This is a INTERVENTIONAL TRANSPLANTATION STUDY WITHOUT DRUGS.
  The INTERVENTION is represented by the INFUSION of DONOR T REGULATORY CELL-ENRICHED LYMPHOCYTES to PATIENTS suffering from REFRACTORY CHRONIC GVHD after ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION.
  The study is single center single arm open label and includes a DOSE ESCALATION phase followed by an EXTENDED PHASE with the MAXIMUM TOLERATED DOSE (MTD).
  During the dose escalation phase each patient will receive three doses of purified donor T reg cells each administered intravenously 1 month apart. Dose levels of purified Tregs will be 5x10e5/kg, 1x10e6/kg and 2x10e6/kg, resulting in three doses of 1.7x10e5/kg, 3.3x10e5/kg and 6.6x10e5/kg, respectively.
  In the dose escalation study at least 9 patients will be required depending on the occurrence of adverse events during the study).
  Patients in the MTD study should be about 10, according to Fleming.
  Interventions: Biological: T reg DLI

INTERVENTIONS:
Biological: T reg DLI — Purified Treg cells will be obtained from the original HSC donor (T reg DLI).
  Tregs preparation will start with unstimulated donor leukapheresis from the original stem cell donor.
  The apheresis product will be provided to the Cell Factory "Calori",Milano, where T reg purification will take place.
  T reg cells will be PURIFIED utilizing the CliniMACS Plus Systems for depletion of CD8 and CD19 positive cells and enrichment for CD25high cells.
  Release Criteria of Treg cell preparation will be defined.
  The product will be infused into the recipient through a venous catheter.
  Other Names: T regulatory cell infusion

SUMMARY:
This is a INTERVENTIONAL TRANSPLANTATION STUDY WITHOUT DRUGS.

The INTERVENTION is represented by the INFUSION of DONOR T REGULATORY CELL-ENRICHED LYMPHOCYTES to PATIENTS suffering from REFRACTORY CHRONIC GVHD after ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION.

The study includes a DOSE ESCALATION PHASE followed by a MTD PHASE as detailed in the following chapter.

The primary objective of the dose escalation study will be SAFETY, leading to the definition of the MTD of T reg cells. For the MTD study the primary objective will be the OVERALL RESPONSE RATE at three months after the 3rd Treg infusion.

The study is single center single arm open label and includes a DOSE ESCALATION phase followed by an EXTENDED PHASE with the MAXIMUM TOLERATED DOSE (MTD).

The aim of the study is to assess whether multiple infusions of donor-derived purified T regulatory cells (T reg DLI) in patients with steroid-refractory chronic GVHD is safe and whether it may induce clinical remission of GVHD.

DETAILED DESCRIPTION:
The procedure under study is the infusion of patients with chronic GVHD with purified Treg cells obtained from the original HSC donor (T reg DLI).

T reg cells are PURIFIED utilizing the CliniMACS Plus Systems for depletion of CD8 and CD19 positive cells and enrichment for CD25high expressing. Treg purification will be performed according to GMP procedure by using the clinical grade CLINI-MACS® device. The protocol is detailed in chapter 3.5

The entire manufacturing process including cell harvesting, transport and Treg purification has been validated.

The feasibility of the selection of nTreg from human peripheral blood using the CliniMACS® System has been previously documented. In these studies, CD8+ and CD19+ cells were undetectable in the final blood products. Final content of CD4+CD25+CD127lo-expressing cells was in mean 79% (range 52-82%) with the improved CD25 enrichment procedure. This protocol has also been validated by two partner Centres in the Treg GENERATION CONSORTIUM, Liège and Boston, with results that meet the release criteria for infusion. These purification procedures provided between 0.98 and 2.93x10e6 Treg per kg. It is noteworthy that the degree of purity in terms of CD4+CD25+CD127- cells ranged between 72.80% and 93.90%.

According to the "Reflection paper on classification of advanced therapy medicinal therapy", published by the Committee for Advanced Therapies (CAT) of the European Medicine Agency on June 20th 2014 [EMA/CAT/600280/2010 Rev.1 lines 118-131] the Treg DLI SHOULD NOT BE CONSIDERED CELL THERAPY MEDICINAL PRODUCTS. Indeed somatic cell therapy medicinal product means a biological medicinal product which fulfils BOTH following two characteristics: (a) contains or consists of cells or tissues that have been subject to substantial manipulation so that biological characteristics, physiological functions or structural properties relevant for the intended clinical use have been altered, or of cells or tissues that are not intended to be used for the same essential function(s) in the recipient and the donor; (b) is presented as having properties for, or is used in or administered to human beings with a view to treating, preventing or diagnosing a disease through the pharmacological, immunological or metabolic action of its cells or tissues. For the purposes of point (a), the manipulations listed in Annex I to Regulation (EC) No 1394/2007, including cutting, grinding, shaping, centrifugation, soaking in antibiotic or antimicrobial solutions, sterilization, irradiation, cell separation, concentration or purification, filtering, lyophilization, freezing, cryopreservation, and vitrification, shall not be considered as substantial manipulations. The procedures listed above for the preparation of the purified T reg product DO NOT FULFILL the definition of substantial manipulation.

Moreover, according to the same document [lines 286-306] T reg DLI SHOULD BE REGARDED as administered for HOMOLOGOUS USE. Indeed, as outlined in "Reflection paper on classification of advanced therapy medicinal therapy" the cells harvested and separated by a simple selection method, and re-administered to fulfil their same essential function will generally be regarded as homologous use. The same essential function for a cell population means that the cells when removed from their original environment in the human body are used to maintain the original function in the same anatomical or histological environment.

Therefore the INFUSION of donor purified T reg cells in TRANSPLANTED PATIENTS (T reg DLI) SHOULD be considered as TRANSPLANTATION rather than the administration of ADVANCED THERAPY MEDICINAL PRODUCT.

The aim of the study is to assess whether multiple infusions of donor-derived purified T regulatory cells (T reg DLI) in patients with steroid-refractory chronic GVHD is safe and whether it may induce clinical remission of GVHD. Based on the observation of the pathophysiological involvement of T regulatory cells in chronic GVHD, the adoptive transfer of donor T regulatory cells appears more reproducible and effective than their in vivo expansion following the administration of drugs.

We will determine feasibility, toxicity and MTD; assess clinical impact and effect on Treg and Tcon homeostasis; and determine whether these effects can be maintained and the extent to which they persist. We will also assess for predictors of response to therapy, both clinical (e.g., patient, disease, concurrent agents) and biological (e.g., degree of Treg expansion; Treg:Tcon ratio; Treg function).

As of 1/1/2015, the current TRIAL PROPOSAL has received funding by the European Union Framework Program on Research and Innovation as a part of a project titled "Repair of tissue and organ damage in refractory chronic graft versus host disease after hematopoietic stem cell transplantation by the infusion of purified allogeneic donor regulatoryT lymphocytes" (acronym TREGeneration, code 643776). The project includes a set of proposals by different European institutions (University of Lisbona, University of Liege, University of Regensburg and the University of Bologna) all investigating the role of Treg DLI in the treatment of chronic GVHD. The GRANT AGREEMENT signed with the EUROPEAN COMMISSION is attached to the proposal.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has undergone allogeneic stem cell transplantation with steroid refractory severe chronic GvHD either occurring post transplant, or induced by donor lymphocyte infusions (DLI) or T-cell add back. The diagnosis of chronic GvHD will based on NIH criteria, 2014 update. Chronic GvHD grading will be performed based on the updated NIH criteria. Severe chronic GVHD will be defined as having SCORE 3 in at least one organ or SCORE 2-3 in the lung.

  * Refractoriness to steroids will be defined based on the following criteria:

    1. use of at least another immunosuppressive medication/strategy besides prophylactic calcineurin inhibitor for previous treatment for cGVHD .
    2. use of prednisone ≥ 0.25 mg/kg/day (or 0.5 mg/kg every other day) (or equivalent dosing of alternate glucocorticoids) for at least 4 weeks prior to enrollment without complete resolution of signs and symptoms.

exclusion criteria:

* Inability to obtain informed consent.
* Patients with documented active EBV, CMV or fungal infection.
* Patients with active HBV, HCV o HIV infection.
* Patients with a diagnosis of solid tumor within the previous year with the exception of NON melanoma skin cancer.
* Patients with evidence of Residual Disease at their last hematologic evaluation.
* Patients in poor clinical conditions (ECOG 3-4)
* Female patients with confirmed pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
OVERALL RESPONSE RATE | 3 months after last T reg infusion
  The response of chronic GVHD to treatment will be assessed per NIH consensus criteria.
  Overall response will be defined as either a complete o partial response.
  Complete Response is defined as resolution of all reversible manifestations related to cGVHD in a specific organ.
  Partial Response will be defined as at least 50% improvement in the scale used to measure disease manifestations related to cGVHD (e.g. a 50% decrease in skin rash from 80% BSA to 40% BSA), in at least one organ or site, without progression in measures at any other organ or site.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Arpinati, Principal Investigator — Hematology and Medical Oncology Institute "L. e A. Seràgnoli"
Locations (1):
- University Hospital St. Orsola-Malpighi Polyclinic, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No